CLINICAL TRIAL: NCT06805682
Title: PEGASE3, Experimental Program of a Standardized Health Protocol Applied to Children Who Benefited from a Child Protection Measure Before the Age of Five: Effectiveness and Efficiency
Brief Title: Prospective Cohort Study of Protected Children
Acronym: ESPER
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Saint-Exupéry Association (Unknown)
Responsible Party: Sponsor
Other Study IDs: APHP230596; PREPS-22-0058 (Other Grant/Funding Number: French Ministry of Health); 2024-A00953-44 (Other: ID RCB)
Record Dates: First submitted 2025-01-17; First posted 2025-02-03 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Mental Health Conditions; Physical Health Status; Child Development
Keywords: Child Protective Services; Child Development; Mental health; Cohort study; Comparative study
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- ESPER: Children under the care of child protective services and followed using usual practices
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Usual Care — Children will be followed using each CPS participating center's usual practices

SUMMARY:
A significant number of children are abused or neglected every year. This exposure is associated with short- and long-term consequences for their mental and somatic health. In France, 308,000 minors are benefiting from at least one child protective service or measure. There are few data on the health status of this population, and how it is evolving. Against this backdrop, interventions are needed to address the many needs of these children early and comprehensively, both in the short and long term.

The PEGASE program, funded by the French government under Article 51, aims to ensure adequate medical follow-up - both somatic and psychiatric - for children taken into care by child protective services (CPS). An evaluation of the program's effectiveness and efficiency is needed to inform public decision-making on the appropriateness of extending it to all children under CPS's care. This requires the creation of a control cohort of children followed by CPS but not benefiting from the PEGASE program, the ESPER cohort (Prospective cohort study of protected children), which will enable us to carry out a comparative evaluation of the PEGASE program, as well as to provide information on the health of children followed by the CPS at the time of their placement and its evolution over time, data which are rare in France.

The main objective is to evaluate the effectiveness of the PEGASE program on the evolution of the mental health of children followed by the CPS after 2 years of follow-up.

DETAILED DESCRIPTION:
A significant number of children are abused or neglected every year. This exposure is associated with short- and long-term consequences for their mental and somatic health, making child abuse a real challenge for society, both on an individual level, in terms of equal opportunities, and on a collective level, from a public health and economic point of view. In France, 308,000 minors benefit from at least one child protection service or measure. There are few data available on the health status of this population and its evolution over time, but they all point to the poor health status of children when first placed into care, with a particularly high prevalence of mental disorders, a low proportion of children benefiting from an initial health check-up, and poor quality of medical follow-up once in care.

In this context, interventions are needed to address early and comprehensively the many needs of children put into care, both in the short and long term. In particular, early detection and reduced delays in the initiation of appropriate medical care appear to have positive long-term effects, reducing medico-social needs. As such, the PEGASE program, which is funded by the French government under Article 51, was developed to ensure adequate medical follow-up - both somatic and psychiatric - for children taken into care by child protective services (CPS).

Children in the PEGASE program are monitored with regular, standardized check-ups, with an initial standardized check-up when the child enters the care facility followed by 20 regular assessments at fixed ages up to the age of 7. Most of these assessments are reinforced in PEGASE by the systematic use of standardized scales to identify potential disorders and developmental delays, so that the necessary care can be implemented at an early stage.

An evaluation of the program's effectiveness and efficiency is needed to inform public decision-making on the appropriateness of extending it to all children in care. As there is no control group in the PEGASE program, this requires the creation of a control cohort of children followed by CPS but not benefiting from the PEGASE program. This is the ESPER cohort (Prospective cohort study of protected children), which will enable us to carry out a comparative evaluation of the PEGASE program, as well as to provide information on the health of children taken into care by the CPS at the time of their placement, and on its evolution over time, data which are rare in France.

The primary objective is to evaluate the effectiveness of the PEGASE program on the evolution of the mental health of children followed by the CPS after 2 years of follow-up.

The secondary objectives are:

* To evaluate the effectiveness of the PEGASE program on the evolution of children followed by the CPS after 1 and 2 years of follow-up, in terms of: mental health, physical health, development (communication, gross motor skills and fine motor skills), care pathway, and school integration,
* To evaluate the cost-effectiveness of the PEGASE program after 2 years of follow-up, and its budgetary impact in the case of generalization,
* To describe the health of children when they are put into care.

An ancillary study is also planned to compare the health of children followed by CPS to the health of children in the general population.

This is a comparative study with an external control group and propensity score matching, calculated from a multivariate logistic regression model that will include a priori: corrected age at inclusion, gender, gestational age, ASQ-SE and ASQ-3 scores at inclusion, reason for placement, current protective measure, and social situation of both parents.

The PEGASE program is already the subject of a separate protocol describing recruitment procedures and follow-up of children benefiting from the program.

The population included in the ESPER study are children taken into care by CPS in 8 volunteer departments not participating in the PEGASE program. They must be aged less than 42 months (i.e. 3 and a half years), arriving for the first time in a participating center, and the holders of parental authority must not object to participation in the study.

The children included the ESPER cohort will be followed as usual by the participating center during the two years of follow-up. Additional data collection by questionnaire will be added to the usual care at inclusion, and then at 1 and 2 years of follow-up either in person or by telephone by the study's local coordinators (if the child is no longer in the facility at the time of collection).

At the inclusion visit, parents or legal guardians will be informed of the study, and their non-opposition will be sought. All socio-demographic, health and school data will be collected by the local coordinators. The ASQ-SE and ASQ-3 questionnaires will be completed, as well as antenatal and pre-placement health data. The data will then be entered into the eCRF by the local coordinators.

At one year of follow-up, the local coordinators will collect health data (from the health records) and school data. If the child is no longer in the facility, data will be collected by telephone from the child's care takers, or from the parents (or holders of parental authority) if the child lives with them. The ASQ-SE and ASQ-3 questionnaires will be completed by the same person. The local coordinators will then enter the data into the tool. The 2-year follow-up visit will be identical to the 1-year visit.

It is planned to include 400 children in the ESPER cohort. The inclusion period is 12 months, and the duration of each child's participation in the study is 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Child under the supervision of child protective services,
* Arriving for the first time in a participating center,
* Less than 42 months old (i.e. 3 and a half years),
* Non-opposition of the holders of parental authority (in the event of impossibility to obtain the non-opposition of both holders of parental authority, the non-opposition of one of them will be obtained).

Exclusion Criteria:

• Children whose child protection measure has not been confirmed by a judicial or administrative decision.

Ages: 0 Months to 42 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children from the control cohort will be included in the participating services of 8 French departments (the territorial level responsible for CPS in France) not participating in the PEGASE program. The child protection measure can be exercised either in an institution, a foster family or an open environment service.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-02-18 (Actual); Primary Completion 2028-02-18 (Estimated); Study Completion 2029-02-18 (Estimated)

PRIMARY OUTCOMES:
Mental health | two years of follow-up
  The primary endpoint is the ASQ-SE questionnaire score after two years of follow-up, dichotomized into: 1/ Failure: the child is above the alert threshold defined for his/her age, indicating the need to initiate or maintain adapted care; 2/ Success: the child is below the age-defined alert threshold (i.e. "within the norm" for his or her age).
  The ASQ-SE assesses socio-emotional development, a reflection of mental health in young children. The higher the score, the more worrying the child's condition.
  As socio-emotional development evolves with age, nine questionnaires are available, depending on the child's age: 2, 6, 12, 18, 24, 30, 36, 48 and 60 months. The questionnaire is made up of around 36 items (the number of items varies according to the age of the child) and is associated with a score (the total score is a function of the number of items, and therefore differs according to age) and alert thresholds.

SECONDARY OUTCOMES:
Mental health_ASQ-SE questionnaire | 1 and 2 years of follow-up
  * Standardized ASQ-SE score: in order to compensate for the variability of the total score scales according to age, the score obtained at the different ages will be standardized between 0 and 100
  * ASQ-SE questionnaire score dichotomized into success or failure
Body mass index | 1 and 2 years of follow-up
  Body mass index will be expressed in z-score, as a function of age and sex
Growth restriction | 1 and 2 years of follow-up
  Percentage of children whose height is below the fifth percentile for their age and sex on a standard growth curve
Communication skills | 1 and 2 years of follow-up
  Assessed with the ASQ-3 "Communication" subscale score. The ASQ-3 screens for developmental delays on five subscales. The lower the score, the more worrying the child's condition. Like the ASQ-SE, the ASQ-3 questions evolve with the child's age, with a maximum score that varies with age, and alert thresholds available for each questionnaire (at 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 27, 30, 33, 36, 42, 48, 54 and 60 months).
  o The score will be dichotomized into failure (score below the alert threshold defined for their age for initiating or maintaining appropriate management) or success (score above the alert threshold), and standardized between 0 and 100 (similarly to the ASQ-SE)
Gross motor development | 1 and 2 years of follow-up
  * Assessed with the ASQ-3 "gross motor skills" subscale score.
  * The score will be both dichotomized as failure or success, and standardized between 0 and 100
Fine motor development | 1 and 2 years of follow-up
  * Assessed with the ASQ-3 "fine motor skills" subscale score.
  * The score will be dichotomized as failure or success, and standardized between 0 and 100
Care pathway | 1 and 2 years of follow-up
  Percentage of children with a complete vaccination protocol
School integration | 1 and 2 years of follow-up
  Number of days of schooling per week
Cost-effectiveness | 2 years of follow-up
  Incremental cost-effectiveness ratio in cost per child below the alert threshold for the ASQ-SE
Costs associated with the generalization of the program | extrapolation at 5 years after hypothetical generalization
  Direct costs associated with children's care and follow-up (healthcare consumption, cost of the PEGASE program…) will be calculated with and without the PEGASE program to assess the budgetary impact of its generalization
Developmental gains associated with the generalization of the program | extrapolation at 5 years after hypothetical generalization
  The number of children with normal development will be calculated with and without the PEGASE program to assess the health gains associated with its generalization
Children's health at admission | measured at study inclusion
  Criteria 1 to 7

OTHER OUTCOMES:
ASQ-3 | at inclusion, 1 year and 2 years of follow-up
  The percentage of children with ASQ-3 questionnaire score dichotomized into success or failure will be compared between ESPER and other existing French children cohorts after matching the cohorts
BMI | at inclusion, 1 year and 2 years of follow-up
  The BMI expressed in z-score, as a function of age and sex will be compared between ESPER and other existing French children cohorts after matching the cohorts
Growth restriction | at inclusion, 1 year and 2 years of follow-up
  The percentage of children whose height is below the fifth percentile for their age and sex on a standard growth curve will be compared between ESPER and other existing French children cohorts after matching the cohorts
Care pathway | at inclusion, 1 year and 2 years of follow-up
  The percentage of children with complete vaccination protocols will be compared between ESPER and other existing French children cohorts after matching the cohorts
School integration | at inclusion, 1 year and 2 years of follow-up
  The number of school days per week will be compared between ESPER and other existing French children cohorts after matching the cohorts

CONTACTS AND LOCATIONS:
Overall Officials: Morgane MICHEL, MD, Principal Investigator — Clinical Epidemiology Unit, Robert Debré Hospital (Assistance Publique - Hôpitaux de Paris)
Locations (8):
- France (8):
  - Maternal and Child Protection - The Eure Department, Évreux, France
  - Departmental institution to support - accompany - educate, Lille, France
  - Moselle Departmental Children's Centre, Metz, France
  - Maternal and Child Protection, Quimper, France
  - Maternal and Child Protection, Rouen, France
  - Maternal and Child Protection, Saint-Brieuc, France
  - Children and Family Home of the Loire, Saint-Genest-Lerpt, France
  - Departmental Observatory for Child Protection, Toulon, France

IPD SHARING:
Plan to Share IPD: No